CLINICAL TRIAL: NCT01072071
Title: The Influence of Furosemide on Fluid Balance and Intra-abdominal Pressure in Mechanically Ventilated Critically Ill Patients With Secondary Intra-abdominal Hypertension
Brief Title: The Influence of Furosemide on Fluid Balance and Intra-abdominal Pressure in Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziekenhuis Netwerk Antwerpen (ZNA) (Other)
Responsible Party: Inneke De laet MD, ZNA Stuivenberg, Intensive Care Unit
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IDL2009/003
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2010-02-22 (Estimated); Status verified 2010-02

CONDITIONS: Intra-Abdominal Hypertension
Keywords: abdominal compartment syndrome; intra-abdominal pressure; furosemide; fluid balance
MeSH Terms: conditions — Intra-Abdominal Hypertension | interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Patients will be receiving standard of care ICU treatment of their underlying disease according to internationally accepted guidelines and recommendations.
- Furosemide group (Experimental): patients will be receiving standard of care ICU treatment of their underlying condition according to international guidelines and recommendations. In addition, furosemide will be administered in continuous infusion as per protocol in order to achieve a preset target diuresis that is adjusted according to haemodynamic tolerance.
  Interventions: Drug: furosemide

INTERVENTIONS:
Drug: furosemide — Loading dose: 0,5mg/kg Start continuous infusion at a dose of 0,1mg/kg/h and titrate according to diuretic response.
  Target value for diuresis = (amount of fluids administered at inclusion/kg/h) + 0.5mL/kg/h If safety check is satisfactory: increase target diuresis with 1mL/kg/h per 4h to a maximum of (amount of fluids administered at inclusion/kg/h) + 2.5mL/kg/h Maximal dose of furosemide: 0.3mg/kg/h Safety check every 4h. Furosemide is administered for 24h. If safety checks are satisfactory, additional periods of 24 can be added up to a maximum of 72h.
  Other Names: Lasix (Sanofi-Aventis)
  Arms: Furosemide group

SUMMARY:
Intra-abdominal hypertension (IAH) is a frequent cause of organ dysfunction in critically ill patients. Secondary IAH is mainly caused by excessive fluid resuscitation.The World Society for the Abdominal Compartment Syndrome (WSACS) recommends using diuretics to remove excess fluids and decrease intra-abdominal pressure (IAP). However, critically ill patients may not tolerate negative fluid balance in the acute phase of their disease and the injured kidney may not respond to diuretics. The aim of this study is to evaluate the influence of furosemide on fluid balance, IAP and kidney function in critically ill patients.

DETAILED DESCRIPTION:
Intra-abdominal hypertension (IAH) and abdominal compartment syndrome (ACS) have been shown to cause organ dysfunction and mortality in different populations of critically ill patients. According to consensus definitions published by the World Society for the Abdominal Compartment Syndrome (WSACS), secondary IAH is due to a disease process outside the abdominal cavity. It is mainly caused by massive fluid resuscitation leading to bowel and abdominal wall edema or increased intra-abdominal volume and decreased abdominal wall compliance. Large observational studies have shown that positive fluid balance is an independent risk factor for mortality. The development of secondary IAH may be one of the mechanisms involved in this phenomenon. This has lead to the hypothesis that prognosis may be improved by managing fluid overload and aiming for a negative fluid balance as soon as possible after the resuscitation phase of the disease.

Several authors have shown in case reports and small series that renal replacement therapy with ultrafiltration can be used successfully to remove excess fluid and lower intra-abdominal pressure (IAP), but renal replacement therapy is invasive and clinicians may be reluctant in considering this therapy in patients with preserved diuresis and kidney function. In an effort to achieve the same goal using a less invasive technique, the new medical management algorithm for IAH published by the WSACS recommends the use of judicious diuresis in order to achieve a negative fluid balance and a decrease in IAP.

However, the kidney is especially sensitive to the deleterious effects of IAH and may be unresponsive to diuretics in the presence of IAH. Also, ongoing inflammation and capillary leak may lead to relative hypovolemia and impaired response to diuretics.

We plan a multicenter study to evaluate the influence of furosemide on fluid balance and IAP in critically ill patients with secondary intra-abdominal hypertension and to document the effect on the function of other organ systems. The aim of this study is to evaluate the feasibility and the safety of the furosemide administration protocol and to provide preliminary data to allow for an adequate power calculation.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18y)
* Sedation (Richmond Agitation and Sedation Score RASS ≤ -3) and mechanical ventilation anticipated to last for at least an additional 72h
* Indication for IAP monitoring according to the recommendations published by the WSACS
* IAP ≥ 12mmHg (intravesical IAP measurement according to WSACS guidelines)
* Absence of surgically treatable abdominal lesions
* Presence of fluid overload

Exclusion Criteria:

* Pregnancy or lactation
* Assisted spontaneous breathing ventilator mode
* Chronic diuretic therapy or on diuretics during inclusion
* Contra-indication to bladder catheterization such as bladder surgery or genitourinary trauma
* Known hypersensitivity to furosemide
* Renal failure Acute Kidney Injury Network (AKIN) class 3
* Patients requiring high dose vasopressors (norepinephrine >0.5µg/kg/min, dobutamine >10µg/kg/min or dopamine>10µg/kg/min, epinephrine>0.5µg/kg/min)
* Intra-abdominal pressure (IAP) >25mmHg at study entry
* DNR orders in effect (other than DNR 1 'no CPR' order)
* Patient not expected to survive for 7 days
* Advanced liver cirrhosis (see pharmaceutical information on furosemide)
* paO2/FiO2 ratio of <100
* oliguria <500mL/24h preceding inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
intra-abdominal pressure | every 4 hours during furosemide administration and daily for 7 days

SECONDARY OUTCOMES:
serum creatinine | daily for 7 days
need for renal replacement therapy | daily for 7 days
ICU mortality | 3 months
acid-base status | daily for 7 days
hospital and 28d mortality | after 28 days and after 6 months
duration of mechanical ventilation | 3 months
ICU length of stay | 3 months
vasopressor dose | daily for 7 days
fluid balance | daily for 7 days
SOFA score | daily for 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- ZNA Stuivenberg Intensive Care Unit, Antwerp, Belgium

REFERENCES:
- See also: World Society for the Abdominal Compartment Syndrome Official Website — http://www.wsacs.org